CLINICAL TRIAL: NCT05776732
Title: Effect of CaviionTM Precaution Medical Adhesive-related Skin Injury in Tumor Patients With PICC Catherizaion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 研2021-0923
Record Dates: First submitted 2023-02-15; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Tumour
Keywords: PICC; medical adhesive-related skin injury
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: 3M CaviionTM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaviionTM group (Experimental): The first nursing is performed within 48 hours after PICC intubation, and each nursing is not more than 7 days thereafter. The nursing contents include skin disinfection, dressing replacement, flushing and locking venous catheters, needleless connector change. After the disinfectant was dried, the experimental group applied CaviionTM on the skin around the catheter and waited for 30 seconds before sticking the dressing.
  Interventions: Other: 3M CaviionTM
- Routine care group (No Intervention): The first nursing is performed within 48 hours after PICC intubation, and each nursing is not more than 7 days thereafter. The nursing contents include skin disinfection, dressing replacement, flushing and locking venous catheters, needleless connector change.

INTERVENTIONS:
Other: 3M CaviionTM — 3M CaviionTM is mainly composed of acrylate trimer, non-toxic, alcohol-free, and compatible with chlorhexidine gluconate and povidone iodine.
  Arms: CaviionTM group

SUMMARY:
Malignant tumor patients are at high risk of medical adhesive-related skin injury（MARSI）.MARSI can cause local skin ulceration, increase the difficulty of fixation and maintenance frequency, even cause unplanned extubation, and increase the pain and economic burden of the patient's re-installation.Malignant tumor patients with long-term PICC are prone to MARSI.CaviionTM can form a protective film on the skin.Applying CaviionTM before using the adhesive can effectively protect the skin and reduce the occurrence of rash.In China, CaviionTM is mostly used in infants and young children, but adults lack corresponding report and application data.Therefore, it is necessary to carry out corresponding randomized controlled study on adult patients, especially malignant tumors

DETAILED DESCRIPTION:
The incidence of medical viscose-related skin injury after PICC intubation is as high as 33.15%. The main types of injury are mechanical injury, moisture-related skin injury, contact dermatitis 8.02%, folliculitis.After radiotherapy and chemotherapy, patients with malignant tumors interfere with the formation of new damaged skin cells.Large doses of immunosuppressive agents further weaken the skin barrier and are prone to skin metabolism and immune function disorder.In this study, patients with malignant tumor after PICC intubation were randomly assigned.The experimental group uses CaviionTM, and the control group does not use CaviionTM. Observe the skin condition one month after the tube placement

ELIGIBILITY:
Inclusion Criteria:

* For malignant tumor patients newly implanted with PICC,indwelling catheter for more than 1 month，Conduct catheter maintenance in my hospital during observation

Exclusion Criteria:

* People with skin disease around PICC tube，Psychopath

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of medical viscose-related skin injury | 1year
  Including mechanical injury (exfoliation, skin tear, tension injury), dermatitis (contact dermatitis and allergic dermatitis), others (immersion and folliculitis)

CONTACTS AND LOCATIONS:
Locations (1):
- 石芸, Hangzhou, ZhwJiang, China

IPD SHARING:
Plan to Share IPD: No